CLINICAL TRIAL: NCT00002441
Title: A Phase III Trial to Determine the Efficacy of Bivalent AIDSVAX B/B Vaccine in Adults at Risk of Sexually Transmitted HIV-1 Infection in North America
Brief Title: Effectiveness of an HIV Vaccine in HIV-Negative Adults in North America Who Are at Risk of HIV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VaxGen (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Prevention
Other Study IDs: VAX 004
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-01

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: HIV-1; Dose-Response Relationship, Drug; Acquired Immunodeficiency Syndrome; AIDS Vaccines; Sexually Transmitted Diseases; Risk Factors; HIV Seronegativity; Antigens, Viral; Alum Compounds
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

INTERVENTIONS:
Biological: MN rgp120/HIV-1 and GNE8 rgp120/HIV-1

SUMMARY:
The purpose of this study is to see if an HIV vaccine, AIDSVAX B/B, can protect adults who are at risk from becoming infected with HIV. Patients who become infected despite immunization will be studied to see if receiving the vaccine before becoming infected will help keep HIV levels (viral load) low.

DETAILED DESCRIPTION:
Volunteers receive 7 blinded, intramuscular vaccinations (at Months 0, 1, 6, 12, 18, 24, 30) containing either the AIDSVAX B/B vaccine or a placebo (aluminum adjuvant only). Volunteers are randomized in a 2 to 1 vaccine-to-placebo ratio. HIV-uninfected persons are followed for a total of 16 visits beginning at screening and continuing until Month 36. Patients who become HIV infected during study are followed every 4 months for at least 24 months.

ELIGIBILITY:
Exclusion Criteria

You will not be eligible for this study if you:

* Use injection drugs.
* Have a history of any serious diseases or conditions, including lymphoma.
* Have ever received an HIV vaccine.
* Have taken post-exposure treatment to prevent HIV infection within 4 weeks prior to study entry.
* Are planning to take other HIV vaccines during this study.
* Are pregnant.
* Have taken certain medications or received certain therapies, including chemotherapy and radiation.
* Have received certain vaccines within 2-4 weeks prior to study entry.

You may be eligible for this study if you:

* Are HIV-negative.
* Are between 18 and 60 years old.
* Are available for 3 years of follow-up.
* Agree to use effective methods of birth control during the study and for 90 days after.
* Are one of the following:
* A woman who is currently in a sexual relationship with an HIV-positive man.
* A woman who has had more than one male partner and at least one sexually transmitted disease (STD) within the past 12 months.
* A man who has sex with men and has had anal intercourse within the past 12 months. (You will not be eligible if you have been in the same relationship with only one HIV-negative man for at least 12 months.)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5000

CONTACTS AND LOCATIONS:
Locations (67):
- United States (63):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Body Positive, Phoenix, Arizona
  - Arizona Clinical Research Ctr Inc, Tucson, Arizona
  - Univ of California / UCI Med Ctr, Orange, California
  - ViRx Inc, Palm Springs, California
  - Univ of California - Davis Med Ctr / CARES, Sacramento, California
  - San Francisco Dept of Hlth / AIDS Office, San Francisco, California
  - San Francisco Gen Hosp, San Francisco, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Santa Clara Public Health Dept, San Jose, California
  - AIDS Research Alliance, West Hollywood, California
  - Denver Hlth and Hosp Authority / Dept of Pub Hlth, Denver, Colorado
  - Johns Hopkins Univ / Ctr for Immun Rsch, Washington D.C., District of Columbia
  - IDC Research Initiative, Altamonte Springs, Florida
  - Community AIDS Resource Inc, Coral Gables, Florida
  - Community AIDS Resource Inc, Fort Lauderdale, Florida
  - Boulevard Comprehensive Care Ctr, Jacksonville, Florida
  - Community AIDS Resource Inc, Riviera Beach, Florida
  - Infectious Disease Research Institute, Tampa, Florida
  - Palm Beach Research Ctr, West Palm Beach, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Univ of Hawaii, Honolulu, Hawaii
  - Chicago Ctr for Clinical Research, Chicago, Illinois
  - Univ of Illinois at Chicago / Dept of Medicine, Chicago, Illinois
  - Howard Brown Health Ctr, Chicago, Illinois
  - Community Hosp Indianapolis, Indianapolis, Indiana
  - Louisiana State Univ Med Ctr / Infect Diseases, New Orleans, Louisiana
  - Fenway Community Health Ctr, Boston, Massachusetts
  - Abbott Northwestern Hosp, Minneapolis, Minnesota
  - Hennepin County Med Ctr, Minneapolis, Minnesota
  - Park Nicollet Med Ctr / Hlth Education, Saint Louis Park, Minnesota
  - St Paul Public Health, Saint Paul, Minnesota
  - Kansas City AIDS Research Consortium, Kansas City, Missouri
  - Saint Louis Univ Hosp / Ctr for Vacc Dev, St Louis, Missouri
  - Wellness Ctr / Las Vegas, Las Vegas, Nevada
  - New Jersey Community Research Initiative, Newark, New Jersey
  - Univ of New Mexico Hlth Sciences Ctr / Dept of Med, Albuquerque, New Mexico
  - Albany Med College / Div of HIV Medicine, Albany, New York
  - AIDS Services Erie County Med Ctr, Buffalo, New York
  - St Luke Roosevelt Hosp, New York, New York
  - New York Univ Med Ctr / Dept of Environmental Med, New York, New York
  - Mount Sinai Med Ctr / Jack Martin Fund Clinic, New York, New York
  - Dutchess County Dept of Health, Poughkeepsie, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - New York Blood Ctr, The Bronx, New York
  - Project Achieve - New York Blood Ctr - Women only, The Bronx, New York
  - Nalle Clinic / Clinical Research Dept, Charlotte, North Carolina
  - PW Clinical Research / LLC, Winston-Salem, North Carolina
  - Case Western Reserve Univ, Cleveland, Ohio
  - Ohio State Univ / ACTU-Univ Clinic, Columbus, Ohio
  - Clinical Pharmaceutical Trials Inc / St Johns Doctors Bldg, Tulsa, Oklahoma
  - Research and Education Group, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Univ of Pittsburgh Med School, Pittsburgh, Pennsylvania
  - Mem Hosp of Rhode Island, Pawtucket, Rhode Island
  - Miriam Hosp, Providence, Rhode Island
  - Omega Med Research, Providence, Rhode Island
  - Nelson Tebedo Health Resource Ctr, Dallas, Texas
  - Oak Lawn Physicians / North TX Ctr for AIDS & Cln Rsch, Dallas, Texas
  - Univ of Texas Med Branch Ctr for Clinical Studies, Galveston, Texas
  - UTMB Ctr for Clinical Studies / St John Prof Bldg, Houston, Texas
  - Univ of Washington, Seattle, Washington
  - Wisconsin AIDS Research Consortium, Milwaukee, Wisconsin
- Canada (2):
  - St Pauls Hosp, Vancouver, British Columbia
  - Ctr Hosp de Universite de Montreal (CHUM), Montreal, Quebec
- Municipal Health Service, Amsterdam, Netherlands
- Clinical Research of Puerto Rico Inc, San Juan, Puerto Rico